CLINICAL TRIAL: NCT05379517
Title: Effects of a Pulmonary Rehabilitation Program (PRP) Versus PRP Plus Pulsed Electromagnetic Field Therapy in Patients With Post-covid Sequelae: A Randomized Clinical Trial Project
Brief Title: Pulmonary Rehabilitation Program With Pulsed Electromagnetic Field Therapy in Patients With Post-covid Sequelae.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Rocío Martín Valero, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMA_RP COVID_2022
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: Covid-19; Pulmonary rehabilitation program; Respiratory rehabilitation; Pulmonary function; Exercise capacity; Pulsed electromagnetic field therapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study is planned as simple blind since the person who performs evaluation is external to participant recruitment and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (No Intervention): Patients in the control group will receive a booklet with general information on a health education program where they will be taught global stretching exercises to be performed themselves at least twice a week at home for 20 minutes. In addition, hygienic postural care will be included.
- Experimental group 1 (Experimental): People will receive a three times-weekly 60 min pulmonary rehabilitation program (PRP) for 8 weeks. Exercise training will be structured in three stages. Exercise will start with a warm-up period (4 minutes); followed by the core phase of aerobic exercises (15-18 minutes), upper and lower limb strength (9 minutes), exercises of the respiratory muscles with diaphragmatic breaths with retentions (10 minutes) and the final cooling-stretching (4 minutes) for a total 45 min, coupled with 15 minutes of breathing retraining with the Threshold Inspiratory Muscle Training® (IMT) device (Philips Respironics). Respiratory muscle training will start at 10% of the initial MIP achieved at startup and will increase by 5% every two weeks until reaching 20% of the initial MIP. The intensity of the exercise training will be at 60-75% of the maximum heart rate rate achieved in the exercise capacity test.
  Interventions: Other: Pulmonary rehabilitation program (PRP)
- Experimental group 2 (Experimental): Patients will receive a pulmonary rehabilitation program (PRP) supplemented with pulsed electromagnetic field therapy. The latter will be applied for 5 weeks, a total of 3 sessions per week. The BTL-6000 Super Inductive System (SIS) will be used with the 'focus field' type manual applicator. The parameters will be: intensity of the magnetic field up to 2.5 Tesla (T), the frequency range to achieve the analgesic effect will vary between 10-20 Hz and, finally, an adjustable relative intensity up to 100%, depending on the perception subjective of the patients. Sessions will last 10 minutes. The parameters and procedure of therapy follow the manufacturer's recommendations. The SIS will be applied in the area where the patient presents the highest level of pain.
  Interventions: Device: Pulsed ectromagnetid field therapy; Other: Pulmonary rehabilitation program (PRP)

INTERVENTIONS:
Device: Pulsed ectromagnetid field therapy — Pulsed electromagnetic field therapy is an innovative therapy. The technology is based on a high intensity electromagnetic field, which positively influences human tissue. It is a form of non-invasive treatment, with good tolerance by patients. High-intensity electromagnetic fields excite neural and muscle cells, which stimulates the human body.
  Arms: Experimental group 2
Other: Pulmonary rehabilitation program (PRP) — This type of physiotherapy program includes: respiratory muscle training, coughing exercises, diaphragmatic training, aerobic training and strength training.
  Arms: Experimental group 1; Experimental group 2

SUMMARY:
Coronavirus 2019 disease can cause important sequelae in the patient, being one of the main affectations of the respiratory system due to bilateral pneumonia and frequently presenting loss of strength, dyspnea, polyneuropathies and multi-organ involvement. Respiratory muscle dysfunction It is one of the most frequent sequelae of this disease. The aim of this study it to assess the effect of pulmonary rehabilitation program (PRP) for 8 weeks vs PRP supplemented with pulsed electromagnetic field therapy (PEFT) vs control group (CG) with health education in people with sequelae of COVID-19 on respiratory capacity and clinical response.

DETAILED DESCRIPTION:
Methods: a single-blind, randomized clinical trial of parallel groups and three branches is presented. Participants will be randomly assigned to the three groups. Thrity-three participants will be randomized assigned either will receive (n=11) PR for 60 minutes, vs (n=11) PR plus PEFT vs (n=11) CG with health education program.

Both groups will receive a three times-weekly 60 min exercise program for 8 weeks. Exercise training will be structured in three stages. Exercise will start with a warm-up period (4 minutes); followed by the core phase of aerobic exercises (15-18 minutes), upper and lower limb strength (9 minutes), exercises of the respiratory muscles with diaphragmatic breaths with retentions (10 minutes) and the final cooling-stretching (4 minutes) for a total 45 min, coupled with 15 minutes of breathing retraining with the Threshold Inspiratory Muscle Training® (IMT) device (Philips Respironics). Respiratory muscle training will start at 10% of the initial MIP achieved at startup and will increase by 5% every two weeks until reaching 20% of the initial MIP. The intensity of the exercise training will be at 60-75% of the maximum heart rate rate achieved in the exercise capacity test. The last group will receive PRP for 8 weeks supplemented with pulsed electromagnetic field therapy (PEFT) three times-weekly 10 min for 5 weeks. Frequency and intensity will be adjusted depending on the perception subjective of the patients.

Before and after the intervention and two months later, the effects on respiratory capacity (spirometry), clinical response, symptoms (pain and dyspnea), respiratory muscle strength, respiratory symptoms, anthropometric, exercise capacity, fatigue, pain will be assessed and quality of life in people with sequelae of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* People between 45 and 65 years old who have overcome COVID-19 and continue with sequelae (fatigue, dyspnea and/or muscle pain) two months after overcoming the illness.
* People with limiting dyspnea of less than grade 2 according to the modified Medical Research Council (mMRC) scale.
* People with diagnostic criteria for COVID-19 according to regulations SEPAR and meet the criteria defined in said regulations for care medical and nursing in a specialized unit (susceptible etiology of specific treatment, who suffered mild-moderate infection and/or repeated exacerbations).

Exclusion Criteria:

* Pregnant people.
* People with pacemakers.
* People who present bleeding.
* People with tumor problems.
* Traumatological, neurological or cardiovascular diseases that prevent patients from performing the training.
* People who present glaucoma, retinal detachment and/or recent cataract surgery.
* People with psychiatric or behavioral disorders condition collaboration with the program.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Forced expiratory volume in the first second of expiration (FEV₁). | Baseline, 8 weeks, 16 weeks.
  Pulmonary function test will be performed using the spirometry equipment Spiro USB MicroMedical® model according to the Guidelines of American Thoracic Society and the European Respiratory Society. Forced expiratory volume in the first second of expiration (FEV₁): volume of air expired during the first second of forced expiration after maximum inspiration. The normal value is ≥ 80%.
Changes in Forced vital capacity (FVC). | Baseline, 8 weeks, 16 weeks.
  Pulmonary function test will be performed using the spirometry equipment Spiro USB MicroMedical® model according to the Guidelines of American Thoracic Society and the European Respiratory Society. Forced vital capacity (FVC): It is expressed as a volume (in ml) and is considered normal when it is greater than 80% of its theoretical value.
Changes in FEV₁ / FVC index. | Baseline, 8 weeks, 16 weeks.
  Pulmonary function test will be performed using the spirometry equipment Spiro USB MicroMedical® model according to the Guidelines of American Thoracic Society and the European Respiratory Society. FEV₁ / FVC index: it is the proportion of the forced vital capacity that an individual exhales in the first second of forced expiration. It must be greater than 75%, although values of up to 70% are accepted.

SECONDARY OUTCOMES:
Changes in Maximal inspiratory pressures (MIP) and maximal expiratory pressures (MEP) | Baseline, 8 weeks, 16 weeks.
  Change in respiratoy muscle function strength will be measured with the MicroRPM® model meter with the participant in sitting. Respiratory pressures will be measured maximum statics following SEPAR recommendations.

OTHER OUTCOMES:
Changes in Body composition | Baseline, 8 weeks, 16 weeks.
  Weight will be measured with a clinical scale (SECA 665, Seca) with a sensitivity of 0.25 k, without shoes, calibrated frequently to 0 g to avoid weight errors. the weight will be expressed in Kg. Height will be calculated with a measuring rod (Holtain Limited) and it will be expressed in m^2. Once the weight and height have been obtained, the BMI will be calculated, which will be expressed in Kg/m^2.
Changes in The Short Performance Physical Battery (SPPB) | Baseline, 8 weeks, 16 weeks.
  Exercise capacity will be evaluated using the "Short Performance Physical Battery" (SPPB). The SPPB is a short physical performance battery that assesses lower extremity function, including balance, strength, and mobility. The SPPB consists of 3 subtests that are walking speed with the 4-meter walk test; the strength and resistance of the lower limbs counting the time required to perform 5 squats "Sit to Stand test" (STS), and the balance standing with the feet together, in tandem and semi-tandem. Each of the subtests is evaluated with a score from 0 to 4. The total score is the sum of the three subtests, obtaining a range from 0 to 12. Higher SPPB scores indicate better physical function.
Changes in The six meter walking test (6-MWT) | Baseline, 8 weeks, 16 weeks.
  Six-meter walking test is a well-established outcome measure in a variety of diseases. It is accurate, reproducible, simple to administer, and well tolerated. The 6MWT is a robust assessment tool for use in clinical trials given its ability to quantitatively evaluate ambulation in a controlled environment.
Changes in Fatigue (Fatigue assessment scale FAS) | Baseline, 8 weeks, 16 weeks.
  Fatigue will be evaluated through the Fatigue assessment scale (FAS). Assess symptoms of chronic fatigue. Total scores can range from 10, indicating the lowest level of fatigue, to 50, indicating the highest level.
Changes in The 36 items Quality of Life Questionnaire | Baseline, 8 weeks, 16 weeks.
  Quality of life will be evaluated through the SF-36 questionnaire. The 36 items of the instrument cover the following scales: Physical function, Physical role, Body pain, General health, Vitality, Social function, Role emotional and mental health. Total scores can range from 0 (worst health status) to 100 (best health status).
Changes in Perception of dyspnea, Medical Research Council (mMRC) | Baseline, through study completion, 16 weeks.
  The perception of dyspnea will be evaluated with the scale of modified Medical Research Council (mMRC) dyspnea. The mMRC is a categorical scale from 0 to 4 points that defines dyspnea among five expressions. The perception of dyspnea will be evaluated with the scale of modified Medical Research Council (mMRC) dyspnea, the measurement will be carried out after performing the 6MWT test.
Changes in Pain, Visual Analogic Scale (VAS) | Baseline, through study completion, 16 weeks.
  Visual Analogic Scale (VAS) is a tool used to help the professional as-sess the intensity of certain sensations and feelings, such as pain. The Visual Analog Scale for pain is composed of a straight line on which an extreme means no pain and the other extreme means the worst pain imaginable.
  Extreme pain corresponds to 10 points. None pain corresponds to 0 points. The patient marks a point on the line that matches the amount of pain they feel. Also known as VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín-Valero, PhD, Study Director — University of Malaga
Locations (1):
- Rocío Martín-Valero, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No